CLINICAL TRIAL: NCT05271032
Title: TRANSPULMONARY TERMODILUTION HEMODYNAMIC PROFILE IN PATIENTS WITH SEPTIC SHOCK AFTER INITIAL RESUSCITATION
Brief Title: PiCCO ASSESSMENT IN PATIENTS WITH SEPTIC SHOCK
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Salvatore Grasso, Director, University of Bari
Other Study IDs: TPTD_CFI01
Record Dates: First submitted 2022-01-20; First posted 2022-03-08 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Septic Patients
  Interventions: Diagnostic Test: use of Trasnpulmonary termodiluetion technique

INTERVENTIONS:
Diagnostic Test: use of Trasnpulmonary termodiluetion technique — All the patients underwent to invasive hemodynamic monitoring through the transpulmonary thermodilution technique (PiCCO, PULSION medical system. Gettinge; Solna, Sweden). Briefly, the technique consists in the administration of a cold saline bolus in superior vena cava while monitoring the corresponding temperature variation through a femoral arterial catheter equipped with a tip thermistor. Accordingly, a 5 French catheter equipped with a tip thermistor was inserted into the femoral artery.
  Other Names: Picco

SUMMARY:
Sepsis is the result of a complex pathological process which involves an intravascular inflammatory state, loss of vascular tone, endothelial injury, extravascular leakage, and often inefficient myocardial contractility. These affect the cardiovascular homeostasis as well as the regional perfusion and tissue oxygenation of patient. The importance of early cardiovascular support in septic patients is the reason why, for about fifteen years, the implementation of standardized resuscitation protocols has been emphasized.

The Surviving Sepsis Campaign Guidelines (SSG) recommend an initial fluid resuscitation followed by use of a vasoactive agent such as norepinephrine for the treatment of patients with septic shock. To understand the impact of the hemodynamic support provided by the resuscitation strategy, the assessment of surrogate clinical parameters is pivotal. According to the current guidelines, the increase of mean arterial pressure (MAP) above 65 mmHg represents the threshold in defining patients as "stable".

Although this strategy has been well established, its impact on the actual hemodynamic profile of the septic patient, remains a subject of ongoing controversy. In this scenario, the transpulmonary thermodilution technique (TPTD) allows invasive assessment of the patient hemodynamic profile in terms of fluid responsiveness, vasomotor status, or global cardiac efficiency. By using this technique, several studies highlighted a wide variability in the individual response of patients undergoing cardiovascular stabilization guided by SSG. This suggests that the implementation of a "customized" resuscitation protocol based TPTD derived parameters rather than resuscitation strategy guided by a fixed mathematic model, could be preferred. However, in daily clinical practice, the use of this advanced hemodynamic monitoring system in not routinely used, though it is often reserved in case of failure of the initial SSG-resuscitation protocol.

The investigators supposed that, even if the initial resuscitative efforts were successful in achieving the SSG targets i.e. by restoring the MAP > 65 mmHg, this could still be inadequate in some patients. Accordingly, the investigators hereby will report the hemodynamic profile of patients with septic shock admitted in ICU.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* admitted in ICU with diagnosis of septic shock

Exclusion Criteria:

* Contraindication at the insertion of the PiCCO catheter; conditions able to bias the transpulmonary thermodilution technique results (atrial fibrillation, extracorporeal membrane oxygenation, valvular disease and/or cardiomyopathy
* Pre-existing respiratory and cardiovascular pathologies
* Pre-existing kidney pathologies

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We enrolled patients admitted in ICU with diagnosis of sepsis shock. Sepsis shock was defined as a probable infectious etiology with sequential organ failure assessment score (SOFA) upper than 2, arterial lactate > 2 mmol dL-1 and contextually hypotension refractory to the initial fluid administration followed by the use of vasoconstrictor agent to sustain the mean arterial pressure (MAP) > 65 mmHg.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
change in Cardiac function index | change from baseline cardiac funziona index (1/min) at 5 hours
  This study aims to assess potential difference in term of cardiac function in septic patient after an initial standardized resuscitation protocol. the cardiac function will be assess thought the PiCCO monitoring system i.e. by assessing the CFI value (1/min).

CONTACTS AND LOCATIONS:
Locations (1):
- Salvatore Grasso, Bari, Italy